CLINICAL TRIAL: NCT02362178
Title: USE OF THROMBOELASTOGRAPHY TO GUIDE BLOOD PRODUCTS REPLACEMENT IN DECOMPENSATED CIRRHOTIC PATIENTS UNDERGOING INVASIVE PROCEDURES
Brief Title: Thromboelastographic Guide for Blood Products in Cirrhotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Lesley De Pietri, Consultant Anaesthestetist, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 133/10
Record Dates: First submitted 2015-01-23; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Liver Cirrhosis; Coagulation Disorder
MeSH Terms: conditions — Liver Cirrhosis; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Thromboelastography (TEG) (Experimental): Patients in the TEG group received fresh frozen plasma at the dose of 10 ml/kg of ideal body weight, only if INR was higher than 1.8 and r time longer than 40 minutes. They received platelets at the amount of 1 apheresis Unit, only if platelets count was lower than 50000/μl and MA was shorter than 30 millimeter.
  Interventions: Procedure: Thromboelastography to guide blood products infusion
- Standard of Care (SOC) (Active Comparator): In the SOC group patients received fresh frozen plasma at the dose of 10 ml/kg of ideal body weight, when INR was higher than 1.8. They received platelets at the amount of 1 apheresis Unit, when platelets count was lower than 50000/μl.
  Interventions: Procedure: Standard of care coagulation tests to guide blood products infusion

INTERVENTIONS:
Procedure: Thromboelastography to guide blood products infusion — A TEG has been performed before invasive procedure and blood products infusion has been decided according to TEG parameters as follow: fresh frozen plasma (FFP 10 ml/kg) in case of r time>40 mm and/or platelets (PLTs 10 units/Kg) for MA<30 mm
  Arms: Thromboelastography (TEG)
Procedure: Standard of care coagulation tests to guide blood products infusion — Patients received FFP (10 ml/kg) if INR>1.8 and/or PLTS (10 units/Kg) If PLTs count < 50000/μl
  Arms: Standard of Care (SOC)

SUMMARY:
Blood products are commonly used before invasive procedures in patients with end-stage liver diseases despite cirrhosis being a thrombophylic state. Traditional coagulation tests (namely INR and PLTs count) are known to be unreliable in predicting bleeding risk before invasive procedures and in representing the real coagulation status of cirrhotic patients. Notwithstanding they are still used to guide blood products administration before invasive procedures. Thromboelastography (TEG) has been shown to be effective in detecting signs of hypo-hypercoagulability possibly being an alternative method to guide blood products transfusion. The aim of this randomized controlled study was to evaluate the efficacy of TEG as a guide for blood products transfusion in cirrhotic patients undergoing invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or imaging-proven liver cirrhosis of any etiology
* INR>1.8 and/or PLTs count <50x103/μl

Exclusion Criteria:

* Ongoing bleeding
* Previous or current thrombotic events defined as any documented blood clot in a venous or arterial vessel
* Ongoing antiplatelet or anticoagulant therapy or stopped less than 7 days before evaluation for the study
* Presence of sepsis according to ACP-SCCP criteria
* Hemodialysis performed within 7 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Comparison in the amount of blood products transfused between the groups | 48 hours from admission
  Comparison of the number of patients receiving blood products (FFPor PLTs or both), and the amount of blood products between the study groups

SECONDARY OUTCOMES:
Post-procedure bleeding | 48 hours from admission
  Comparison of the number of patients having bleeding episodes after procedure between the study groups
Survival | 90 days patient survival
  Comparison of patients survival between the study groups
Transfusion related side effects | 48 hours from admission
  Comparison of the number of patients presenting transfusion side effects between the study groups
Procedure-related complications | during hospitalization (mean 4 weeks)
  Comparison of the number of patients presenting post-procedures complication other than bleeding between the study groups
Comparison between blood products costs between groups | 48 hours from admission

CONTACTS AND LOCATIONS:
Overall Officials: Lesley De pietri, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena-Policlinico, Division of Anaesthesiology and Intensive Care Unit